CLINICAL TRIAL: NCT06753214
Title: Effectiveness of Telemedicine-Based Education for Caregivers on Asthma Control in Children With Uncontrolled Asthma: A Randomized Controlled Trial
Brief Title: Telemedicine Education for Caregivers and Asthma Control in Children
Acronym: TCARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Can Tho University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Ly Cong Tran, Lecturer, Can Tho University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2313/QD-DHYDCT; U1111-1317-1148 (Other: The Universal Trial Number (UTN))
Record Dates: First submitted 2024-12-22; First posted 2024-12-31 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Uncontrolled Asthma; Telemedicine-Based Education
Keywords: Asthma; Pediatrics; Telemedicine; Uncontrolled asthma
MeSH Terms: conditions — Asthma | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard care (Sham Comparator): The caregivers will receive a video call from the intervention researcher shortly for a health check and a reminder to follow the scheduled appointments.
  Interventions: Other: Standard Care (in control arm)
- Telemedicine (Experimental): Caregivers in the intervention group will receive a video call from the intervention researcher within 15 minutes. The call will include education on avoiding factors related to uncontrolled asthma, reminders about treatment adherence, and following the scheduled appointments. Caregivers will be shown a visual demonstration of proper inhaler use, and they can ask questions about the video's practical steps at any time during the conversation. Additionally, questions about asthma management will be discussed, and tailored advice will be provided according to each child's condition.
  Interventions: Other: Telemedicine-Based Education

INTERVENTIONS:
Other: Telemedicine-Based Education — Intervention through telemedicine
  Arms: Telemedicine
Other: Standard Care (in control arm) — Sham comparator through telemedicine
  Arms: Standard care

SUMMARY:
Asthma control in pediatric patients remains a critical issue for healthcare providers. Telemedicine has emerged as an effective solution for overcoming distance barriers in healthcare delivery. This study aims to utilize telemedicine-based education for caregivers to improve asthma control in children with uncontrolled asthma. By providing remote guidance and support, the study seeks to enhance caregivers' knowledge and management practices, ultimately leading to better asthma outcomes for pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric asthma patients diagnosed according to the GINA guidelines, classified as having uncontrolled asthma, are managed and followed up for at least 1 month at the pediatric asthma unit of the outpatient department.

Exclusion Criteria:

* Pediatric patients who do not cooperate or are unable to complete the Childhood Asthma Control Test questionnaire.
* Caregivers who cannot complete the questionnaires related to the assessment of asthma control and associated factors.
* Pediatric patients who have siblings participating in the study.
* Patients currently participating in another clinical study (excluding non-interventional studies or registries).
* Failure to return for a second visit within 6 months following enrollment.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The improvement of asthma control | At second follow-up visit (ranging from 4 to 24 weeks after enrollment)
  The patients will be evaluated for asthma control using the Childhood Asthma Control Test (C-ACT) for children aged 4-11 or Asthma Control Test (ACT) for children aged 12 and older. This evaluation will also be compared to the baseline to determine whether there is improvement after the intervention period.

SECONDARY OUTCOMES:
The improvement of caregiver's knowledge regarding asthma control | At second follow-up visit (ranging from 4 to 24 weeks after enrollment)
  The caregiver's knowledge regarding asthma will be assessed using a validated questionnaire. This evaluation will also be compared to the baseline to determine whether there is improvement after the intervention period.
The improvement of caregiver's attitudes toward asthma management | At second follow-up visit (ranging from 4 to 24 weeks after enrollment)
  Caregiver's attitudes toward asthma management will be assessed using a set of questions designed to evaluate their perspectives on key aspects of asthma care, including the importance of regular doctor visits, adherence to controller medications, following prescription instructions, proper cleaning of inhaler devices, and mouth rinsing after inhaler use. The evaluation will be compared to baseline data to determine whether there is an improvement in caregivers' attitudes after the intervention period.
The improvement of proper inhaler technique usage | At second follow-up visit (ranging from 4 to 24 weeks after enrollment)
  The patients will be evaluated on their proper inhaler use technique using a consistent checklist. This evaluation will be compared to the baseline to determine whether there is any improvement after the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Nghia Quang Bui, MD, PhD, Study Chair — Can Tho University of Medicine and Pharmacy; Ly Cong Tran, MD, MSc, Study Director — Can Tho University of Medicine and Pharmacy; Thang Hoang Le, MD, Principal Investigator — Can Tho University of Medicine and Pharmacy
Locations (1):
- Can Tho Children's Hospital, Can Tho, Vietnam

IPD SHARING:
Plan to Share IPD: No
Prohibited from regulations and contracts; Fear of inappropriate use of data